CLINICAL TRIAL: NCT00333437
Title: Pulmonary Involvement in Scleroderma: Safety and Efficacy of Mycophenolate Mofetil in Scleroderma Patients
Brief Title: Pulmonary Involvement in Scleroderma: A Clinical Study of the Safety and Efficacy of Mycophenolate Mofetil in Scleroderma Patients With Lung Involvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEL371
Record Dates: First submitted 2006-06-02; First posted 2006-06-05 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-09

CONDITIONS: Scleroderma, Systemic
Keywords: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Mycophenolate Mofetil
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Mycophenolate mofetil

SUMMARY:
Researchers from the Division of Pulmonary and Critical Care Medicine at University of California, San Francisco (UCSF) are conducting a study to evaluate whether mycophenolate mofetil (an immunosuppressive medication, trade named CellCept) is safe and effective for preventing the lung damage from scleroderma from getting worse.

DETAILED DESCRIPTION:
The proposed study is designed to evaluate the safety and efficacy of mycophenolate mofetil (CellCept) for the treatment of symptomatic pulmonary alveolitis due to systemic sclerosis (SSc). This study utilizes a prospective, open-label, experimental design.

Primary Hypothesis: The alveolitis in patients with SSc, as defined by decreased forced vital capacity (FVC), bronchoalveolar lavage (BAL), and High Resolution Chest Tomography (HRCT) is responsive to 1 year of daily mycophenolate mofetil therapy.

Secondary Hypothesis: Quality of life, six-minute walk and single-breath diffusing capacity for carbon monoxide (DLCO) improve in patients with SSc mediated alveolitis after therapy with mycophenolate mofetil. This response to therapy is associated with a change in the inflammatory cytokine profile present in BAL fluid.

ELIGIBILITY:
Inclusion Criteria:

* To participate in this study, patients must first undergo a BAL and HRCT. To be eligible to undergo HRCT and BAL (under the purview of this trial), prospective patients must meet the following criteria:

  * Aged 21-70.
  * Negative pregnancy test (with a sensitivity of at least 50 mIU/mL) for females of child-bearing potential
  * All patients must fulfill the criteria for SSc by American College of Rheumatology (ACR) criteria (Subcommittee for Scleroderma Criteria 1980).
  * FVC < 85% of predicted.
  * SSc for no more than 7 years with onset defined as the date of the first non-Raynaud manifestation.
  * Patients may have limited (cutaneous thickening distal but not proximal to elbows and knees, with or without facial involvement) or diffuse (cutaneous thickening proximal to elbows and knees, often involving the chest or abdomen) cutaneous SSc (Medsger 1995).
  * Abnormal DLCO and abnormalities on the plain chest radiograph are not required, although a normal DLCO would be unusual in the face of significant ventilatory restriction due to SSc lung disease.
* To be eligible to take study medication, the patient must meet not only the criteria above, but also must have ≥ 3.0% neutrophils or ≥ 2.0% eosinophils in screening BAL fluid and/or ground glass opacification on HRCT.
* Women of childbearing potential should have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 1 week before beginning therapy. CellCept therapy will not be initiated until a report of a negative pregnancy test has been obtained.
* Effective contraception must be used before beginning CellCept therapy, during therapy, and for 6 weeks following discontinuation of therapy, even where there has been a history of infertility, unless due to hysterectomy. Two reliable forms of contraception must be used simultaneously unless abstinence is the chosen method. If pregnancy does occur during treatment, the physician and patient should discuss the desirability of continuing the pregnancy.

Exclusion Criteria:

* FVC < 45% of predicted or DLCO (corrected for hemoglobin [Hgb] but not for alveolar volume) < 35% of predicted (suggestive of severe, probably irreparable, disease).
* Leukopenia (white blood cell count < 4000) or thrombocytopenia (platelet count < 100,000).
* Serum creatinine ≥ 2.0 mg/dl.
* Pregnancy, breast feeding, unreliability, drug abuse, or chronic debilitating disease.
* Uncontrolled congestive heart failure.
* Active infection of the lung, or elsewhere, whose management would be compromised by mycophenolate mofetil.
* Prior treatment for alveolitis with mycophenolate mofetil or prior or current treatment for alveolitis with: D-penicillamine, methotrexate, colchicine, Potaba, or azathioprine.
* Other serious concomitant medical illness (e.g., cancer).
* Forced expiratory volume in 1 second (FEV1)/FVC ratio < 65%.
* If of childbearing potential, failure regularly to be employing two reliable means of contraception (i.e., condom, abstinence, intrauterine device (IUD), tubal ligation, vasectomy)
* Pulmonary hypertension (defined as an estimated systolic blood pressure (SBP) ≥ 35 mmHg measured by echocardiogram).
* Smoking of cigars, pipes, or cigarettes during the past 6 months.
* Clinically significant abnormalities on chest x-ray or HRCT scan other than interstitial lung disease (e.g., lung mass, evidence of active pulmonary infection).
* Use of prednisone (or equivalent) in doses > 10 mg per day.
* Does not have ≥ 3.0% neutrophils or ≥ 2.0% eosinophils on screening BAL fluid and does not have ground glass opacification on HRCT.
* Unable to take oral medication.
* Not able to comply with study procedures in the opinion of the investigator.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Golden, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, 400 Parnassus Ave, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 patients were screened at one clinical site (UCSF) in the United States
Pre-assignment Details: One patient screened for enrollment did not meet eligibility criteria
Groups:
- Single-group Study Treatment: Study subjects receive standard mycophenolate dosing 2 grams/day.
Period: Overall Study
Arm/Group | Single-group Study Treatment
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Study subjects receive standard mycophenolate dosing.
Arm/Group | Treatment
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 52.57 (7.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Forced Vital Capacity (FVC)
Description: compare pre- and post-therapy FVC (post- minus pre-). Forced vital capacity (FVC) is the volume of air (liters) that can forcibly be blown out after full inspiration.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Treatment
Number analyzed (Participants) | 7
Liters | 0.1786 (0.1613)
Statistical Analysis 1: Comparison: Treatment; H(0): post-pre FVC (liters) = 0; Test type: Superiority or Other; p = 0.026, t-test, 2 sided — Not adjusted; Change from Baseline = 0.1786, 95% CI 2-sided [0.0294 to 0.3277], Standard Deviation 0.1613

2. Secondary Outcome: Mean Change in Bronchoalveolar Lavage (BAL) Components (Neutrophils, Eosinophils)
Description: BAL samples were colleected from the affected lobe (as determined by lung CT scans) before beginning and after completing study therapy.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: Cells/uL
Groups:
- Treatment: Study subjects receive standard mycophenolate dosing 2 grams/day.
Arm/Group | Treatment
Number analyzed (Participants) | 7
Cells/uL
  Mean change in neutrophil count | -3 (8.1)
  Mean change in eosinophil count | -6.3 (16.4)
Statistical Analysis 1: Comparison: Treatment; H(0): Post-pre neutrophil count = 0; Test type: Superiority or Other; p = 0.3652, t-test, 2 sided — significant p<0.05; Mean Difference (Final Values) = -3, 95% CI 2-sided [-10.49 to 4.4945], Standard Deviation 8.1035
Statistical Analysis 2: Comparison: Treatment; H(0): post-pre eosinophil count = 0; Test type: Superiority or Other; p = 0.3485, t-test, 2 sided — significant p<0.05; Mean Difference (Final Values) = -6.286, 95% CI 2-sided [-21.41 to 8.8426], Standard Deviation 16.358

3. Secondary Outcome: Change in Shortness of Breath (Self-reported)
Description: Participants reported frequency of shortness of breath experienced with exertion
Time Frame: Baseline, 12 months
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 7
participants
  Patient-reported less shortness of breath | 6
  Patient-reported no change in shortness of breath | 1
  Patient-reported increased shortness of breath | 0

4. Secondary Outcome: Mean Change in Six Minute Walk Distance
Description: Comparison of 6-minute walk distance before beginning and after completing study therapy
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Treatment
Number analyzed (Participants) | 7
Feet | 264.3 (194.7)
Statistical Analysis 1: Comparison: Treatment; H(0): post-pre walk distance = 0; Test type: Superiority or Other; p = 0.0115, t-test, 2 sided — Significant p<0.05; Not adjusted; Mean Difference (Final Values) = 264.26, 95% CI 2-sided [84.256 to 444.32], Standard Deviation 194.66

5. Secondary Outcome: Mean Change in Diffusion Capacity of the Lung for Carbon Monoxide (DLCO)
Description: DLCO was measured before beginning and after completion of study therapy
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Treatment
Number analyzed (Participants) | 7
Liters | 1.86 (1.50)
Statistical Analysis 1: Comparison: Treatment; H(0): Post-pre DLCO = 0; Test type: Superiority or Other; p = 0.0167, t-test, 2 sided — significant p<0.05; Mean Difference (Net) = 1.8643, 95% CI 2-sided [0.4758 to 3.2527], Standard Deviation 1.5013

ADVERSE EVENTS:
Time Frame: 12 months
Description: Appropriate safety and serological studies were obtained prior to starting study medication and on a regular basis throughout the study. Patients were asked to keep a diary of significant medical events occurring between visits.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=7)
Leukopenia (Blood and lymphatic system disorders) | 1 (7) — Patient was hospitalized
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=7)
Gastrointestinal distress (Gastrointestinal disorders) | 1 (1) — Patient was unable to tolerate full dose of study drug because of GI distress

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes